CLINICAL TRIAL: NCT03646097
Title: Impact of Real-time Angiographic Co-registered OCT on PCI Results - the Randomized OPTICO-integration II Study
Brief Title: Impact of Real-time Angiographic Co-registered OCT on PCI Results - the OPTICO-integration II Study
Acronym: Integration-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, David Manuel Leistner, PD Dr. med., Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPTICO-Integration II
Record Dates: First submitted 2018-08-05; First posted 2018-08-24 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Ischaemic Heart Disease
Keywords: OCT; Co-Registration; Stent; PCI; Geographical mismatch; Edge Dissection
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blinded-group (Active Comparator): Lesion assessment, selection of PCI landing zone as well as stent selection will be performed by investigators only based on angiographic lesion evaluation (standard care)
  Interventions: Procedure: Angio-PCI
- OCT-group (Active Comparator): Patients underwent OCT-imaging before PCI. Lesion assessment, selection of PCI landing zone as well as stent selection will be performed by investigators based on OCT findings
  Interventions: Procedure: OCT-PCI
- ACR-group (Experimental): Patients underwent ACR-imaging before PCI. Lesion assessment, selection of PCI landing zone as well as stent selection will be performed by investigators based on ACR-findings
  Interventions: Procedure: ACR-PCI

INTERVENTIONS:
Procedure: Angio-PCI — PCI only with angiography and without OCT findings
  Arms: Blinded-group
Procedure: OCT-PCI — PCI with OCT-measurements but no transfer of landingzone-markers to angiography
  Arms: OCT-group
Procedure: ACR-PCI — PCI with OCT-measurements and transfer of landingzone-markers to angiography
  Arms: ACR-group

SUMMARY:
Intracoronary optical coherence tomography (OCT) imaging allows for high-resolution characterization of coronary lesions. Difficulties in matching cross-sectional OCT-images with angiographic lesion localization, however, may limit its clinical utilization. The investigators sought to prospectively assess the impact of a novel system of real-time OCT-coregistration with angiography (ACR) compared to OCT alone and to the clinical standard proceeding (angiographic guided-PCI) all used for coronary lesion evaluation before percutaneous coronary interventions (PCI). The investigators hypothesize that the use of ACR will lead to less incidence of insufficient covered coronary lesions (geographical mismatch) and/or a less rate of edge dissections after PCI (combined primary study endpoint)

DETAILED DESCRIPTION:
In this randomized blinded pilot-study the effect of pre-PCI planning by angiographic-co-registered OCT (ACR) compared to OCT or angiographic evaluation alone with respect to the entire result after PCI will be investigated. A special focus (primary endpoint) will be on the incidence of geographical mismatch (GM) and/or major edge dissections. Eligible patients will be randomized in three groups.

Group 1 Pre-PCI-OCT: Patients underwent OCT-imaging before PCI. Lesion assessment, selection of PCI landing zone as well as stent selection will be performed by investigators based on OCT findings.

Group 2: Pre-PCI-ACR: Patients underwent ACR-imaging before PCI. Lesion assessment, selection of PCI landing zone as well as stent selection will be performed by investigators based on ACR-findings.

Group 3:OCT-Blinded/Angiographic guided PCI: Lesion assessment, selection of PCI landing zone as well as stent selection will be performed by investigators only based on angiographic lesion evaluation (standard care).

For outcome analysis all study groups underwent post-PCI-OCT imaging as soon as investigators assume angiographic justiciable PCI-results (TIMI III, no residual stenosis > 50%; no angiographic definable or suspicious edge dissections, angiographic acceptable stent expansion without evidence for malapposition). OCT imaging analysis will be performed within a OCT core-lab by two investigators blinded for the randomization group.

ELIGIBILITY:
Inclusion Criteria:

* Patient with indication for coronary angiography for angina (stable or unstable), silent ischemia (a visually estimated target lesion diameter stenosis of ≥70%, a positive invasive or non-invasive test must be present), or NSTE-ACS
* male or non pregnant female patient
* Signed written informed consent

Exclusion Criteria:

* Known neoplasia on treatment / without a curative therapeutic approach
* Presence of one or more co-morbidities which reduces life expectancy to less than 24 months
* Estimated creatinine clearance <40 ml/min
* Cardiogenic shock
* Hemodynamic instability because of arrhythmia
* Known left ventricular ejection fraction (LVEF) <30%.
* Therapy requiring psychiatric disorder
* Patient is participating in any other investigational drug or device clinical trial that has not reached its primary endpoint.
* Women who are pregnant or breastfeeding
* Refusal of study participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of a combined endpoint based on "major edge dissections" (I) AND/OR "geographical mismatch" (II) [%] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Analysis of primary endpoint will be assessed by evaluation of proximal and/or distal stent end.
  I) Major edge dissection (MED):
  Major: ≥60 degrees of the circumference of the vessel at site of dissection and/or ≥3 mm in length
  II) Geographical mismatch (GM):
  Untreated plaque with a minimal lumen area <4,5mm2 within 5mm of the reference segment.
  In the postPCI-OCT analysis it is considered as no geographical mismatch, if:
  1. the segment of the lesion is fully covered AND
  2. the stent protrudes maximal 5mm beyond the predetermined landing zone.
  If one of these criteria is not fulfilled, it is considered as geographical mismatch

SECONDARY OUTCOMES:
Incidence of "major edge dissections" [%] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  All secondary endpoints of OCT will be assessed by evaluation of proximal and/or distal stent end/segment.
Incidence of "all edge dissections" (major (I) and minor (II)) [%] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  (I) ≥60 degrees of the circumference of the vessel at site of dissection and/or ≥3 mm in length (II) Any visible edge dissection <60 degrees of the circumference of the vessel and < 3 mm in length
Incidence of "geographical mismatch" [%] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  see primary endpoint
Stent expansion [%] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Defined by the MSA achieved relative to the proximal or distal reference segments.
  The stent length is divided into 2 equal segments (proximal and distal), and the MSA is determined in each segment.
  * Optimal stent expansion: The MSA of the segment is ≥95% of the related reference lumen area
  * Acceptable stent expansion: The MSA of the segment is ≥90% and <95% of the related reference lumen area
  * Unacceptable stent expansion: The MSA of the segment is <90% of the related lumen area
Inacceptable stent expansion [%] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  see outcome 5
Incidence of "malapposition" [%] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Incompletely apposed stent struts in at least 5 consecutive OCT-frames (defined as stent struts clearly separated from the vessel wall (lumen border/plaque border) without any tissue behind the struts with a distance from the adjacent intima of ≥0.2 mm and not associated with any side branch).
  Malapposition will be further classified as:
  A) Major: If associated with stent underexpansion (unacceptable stent expansion as defined above) B) Minor: If not associated with significant underexpansion (optimal or acceptable stent expansion as defined above) C) Major and minor
Distance between target and actual lesion coverage [mm] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Defined as the distance between target landing zone and actual landing zone of stent location (proximal and distal end). Therefore, the lesion is divided in two equal halves, so that every segment (proximal and distal) can be analyzed for itself.
Minimal Stent Area (MSA) of target lesion [%] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Minimal lumen area covered by stent.
Acute Luminal Gain of target lesion [mm] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Gain of Minimal Lumen Diameter (MLD) between prePCI- and postPCI-OCT
Procedure time [min] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Time from reaching the ostium with the guide catheter until pullback of the last one.
Total fluoroscopy time [min] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Total time required for diagnostic angiography and PCI.
Total contrast volume [ml] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Total amount of contrast used for entire intervention (including OCT-pullbacks)
Total stent length [mm] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Addition of each stent length which were used for target lesion
Total number of stents | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Number of stents which were used for target lesion
Maximal stent diameter [mm] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Maximal stent diameter used for target lesion
Complications associated with OCT-examination [%] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Complications between advancing and pullback of OCT catheter
Complications during hospitalization [%] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Defined as: new ACS; stent thrombosis of study culprit lesion; new unplaned coronary angiography; new revascularization (PCI/CABG); apoplex/TIA; pacemaker implantation; anaphylactic shock; contrast-induced nephropathy; bleeding; death
DOCE within target lesion [%] | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Device-oriented composite endpoint within the target lesion. Defined as cardiovascular death, myocardial infarction OR target-lesion revascularization. This composite endpoint will be checked during a follow up after 1 and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: David M Leistner, PD Dr. med., Principal Investigator — Managing Senior Physician
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided